CLINICAL TRIAL: NCT00844636
Title: A Randomized Trial of Blunt Needles for the Reduction of Needlestick Injuries During Cesarean Section
Brief Title: A Trial of Blunt Needles for the Reduction of Needlestick Injuries During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Bridget Williamson MD, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Blunt Needles - Cesarean
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Glove Perforations; Needlestick Injuries
Keywords: Needlestick injuries; Glove perforations; Blunt Needles; Glove perforations of surgeons, assistants; Needlestick injuries of same
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sharp Needles (Active Comparator): Sharp needles to close uterus, fascia and skin during cesarean section
  Interventions: Device: Sharp needle
- Blunt Needles (Active Comparator): Assignment to blunt needles to close uterus, fascia and skin during cesarean section
  Interventions: Device: Blunt needles

INTERVENTIONS:
Device: Sharp needle
  Arms: Sharp Needles
Device: Blunt needles
  Arms: Blunt Needles

SUMMARY:
The objective of this study was to determine if blunt needle use during cesarean section closure protects against glove perforation and percutaneous injury to the surgeon and surgical assistant. A secondary objective was to determine physician satisfaction with blunt needles during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Pregnant
* Undergoing a cesarean section

Exclusion Criteria:

* Under age 18
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number of observed glove perforations | 1 day
  review post-op

SECONDARY OUTCOMES:
Physician satisfaction with the needle assignment | 1 day
  Rating scale 1-5 (1 being least satisfied and 5 being very satisfied); review post-op

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sullivan, MD, Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Sullivan S, Williamson B, Wilson LK, Korte JE, Soper D. Blunt needles for the reduction of needlestick injuries during cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2009 Aug;114(2 Pt 1):211-216. doi: 10.1097/AOG.0b013e3181ae9b4a. PMID 19622979